CLINICAL TRIAL: NCT00499018
Title: A Randomised Multicentric Phase III Study for the Treatment of Young Patients With High Risk (IPI 2-3) Diffuse Large B-Cell Lymphoma. Dose Dense Chemotherapy + Rituximab +/- Intensified High Dose Chemoimmunotherapy With Support of Peripheral Autologous Stem Cells.
Brief Title: Dose Dense Chemotherapy + Rituximab +/-Intensified High Dose Chemoimmunotherapy With Support of Peripheral Autologous Stem Cell in Diffuse Large B-Cell Lymphoma
Acronym: DLCL04
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Umberto Vitolo, A.O. San Giovanni Battista - Molinette Torino
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIL-DLCL04; EudraCT number 2007-000275-42
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Diffuse Large B-Cell Lymphoma; IPI≥2
Keywords: Large B-Cell Lymphoma; Rituximab; Autologous Stem Cell Transplantation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; pegfilgrastim; Mitoxantrone; Cytarabine; Lenograstim; Carmustine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): R-MegaCHOP14 x 4 Restaging + R-MAD + MAD + BEAM + ASCT
  Interventions: Drug: Rituximab; Drug: Ciclofosfamide; Drug: Doxorubicina; Drug: Vincristina; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Mitoxantrone; Drug: ARA-C; Drug: Lenograstim; Drug: BCNU; Drug: VP-16; Procedure: ASCT
- 1 BIS (Experimental): R-CHOP14 x 4 Restaging + R-MAD + MAD + BEAM + ASCT
  Interventions: Drug: Rituximab; Drug: Vincristina; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Lenograstim; Drug: BCNU; Drug: ARA-C; Drug: VP-16; Procedure: ASCT; Drug: Ciclofosfamide; Drug: Doxorubicina
- 2 (Experimental): R-MegaCHOP14 x 4 Restaging + R-MegaCHOP x 2
  Interventions: Drug: Rituximab; Drug: Ciclofosfamide; Drug: Doxorubicina; Drug: Vincristina; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Mitoxantrone; Drug: ARA-C
- 2 BIS (Experimental): R-CHOP14 x 4 Restaging + R-CHOP14 x 4
  Interventions: Drug: Rituximab; Drug: Vincristina; Drug: Prednisone; Drug: Ciclofosfamide; Drug: Doxorubicina

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 day 1
Drug: Ciclofosfamide — 1200 mg/m2 day 1
  Arms: 1; 2
Drug: Doxorubicina — 70 mg/m2 day 1
  Arms: 1; 2
Drug: Vincristina — 1,4 mg/m2 (max 2 mg) day 1
Drug: Prednisone — 100 mg day g 1-5
Drug: Pegfilgrastim — 6 mg day +1
  Arms: 1; 1 BIS; 2
Drug: Mitoxantrone — 8 mg/m2/days 1-3
  Arms: 1; 2
Drug: ARA-C — 2000 mg/m2/12h day 1 - 3
  Arms: 1; 2
Drug: Lenograstim — 5 μg/Kg/days +2
  Arms: 1; 1 BIS
Drug: BCNU — 300 mg/m2 day -7
  Arms: 1; 1 BIS
Drug: ARA-C — 200 mg/m2/12 days -6,-5,-4,-3
  Arms: 1; 1 BIS
Drug: VP-16 — 100 mg/m2/12h days -6,-5,-4,-3
  Arms: 1; 1 BIS
Procedure: ASCT — PBSC Reinfusion
  Arms: 1; 1 BIS
Drug: Ciclofosfamide — 750 mg/m2 day 1
  Arms: 1 BIS; 2 BIS
Drug: Doxorubicina — 50 mg/m2 day 1
  Arms: 1 BIS; 2 BIS
Drug: Vincristina — 1,4 mg/m2 (max 2 mg) day 1
  Arms: 1 BIS; 2 BIS

SUMMARY:
The purpose of this study is to define an improvement in patients randomized in four different arms:

Arm 1: R-MegaCHOP14x4 + R-MAD + MAD + BEAM + ASCT; Arm 1BIS: R-CHOP14x4 + R-MAD + MAD + BEAM + ASCT; Arm 2: R-MegaCHOP14x4 + R-MegaCHOP14x2; Arm 2BIS: R-CHOP14x4 + R-CHOP14x4; Which are different in dose dense chemotherapy + Rituximab with or without intensified high dose chemoimmunotherapy and support of peripheral autologous stem cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60;
2. Histological confirmed diagnosis of Diffuse Large B-Cell Lymphoma CD20+ (newly diagnosis or shifted from low grade NHL and not previously treated) or of Follicular Lymphoma grade III according to REAL/WHO Classification.
3. Advanced stage II, stage III and stage IV with at least two aa-IPI risk factors.
4. Age-adjusted IPI 2-3.
5. ECOG performance status 0-2.
6. LVEF>45%, measured with echocardiography.
7. Normal hepatic, renal and pulmonary functions.
8. HIV, HCV and HBV negativity.
9. HCV+ admitted only in histologically confirmed absence of replication marks.
10. Positive serology for HBV (occult carriers: AntiHBcAg+, HbsAg-, AntiHBsAg+/-) admitted only upon negativity of weakly positive HBV-DNA test.
11. Life expectancy > 3 months.
12. Negative pregnancy test.
13. Written Informed Consent.

Exclusion Criteria:

1. Histological diagnosis of:

   * Lymphoblastic NHL
   * Burkitt's Lymphoma
   * CD 20 negative B-cell Lymphoma
   * grade I-IIIa Follicular Lymphoma
   * Mantle Cell Lymphoma
   * Primary mediastinal NHL with exclusively intrathoracic localization.
2. Age > 60
3. Stage I disease
4. Age-adjusted IPI 0-1
5. ECOG-PS>3, if not related to Lymphoma
6. Renal impairment (creatinine>1,2 mg/dl or creatinine clearance < 60ml/min)
7. Hepatic impairment (AST/ALT or bilirubin > 2,5 times normal limit, unless due to Lymphoma)
8. HIV positive patients and/or with HBV or HCV active infection(documented by HBV-DNA and HCV-RNA positive tests)
9. Clinically significant secondary cardiovascular disease e.g. uncontrolled hypertension (resting diastolic blood pressure > 115 mmHG), uncontrolled multifocal cardiac arrhythmias, symptomatic angina pectoris or congestive cardiac failure NYHA class III-IV
10. LFEV<45%
11. Severe diabetes mellitus difficult to control with adequate insulin therapy
12. Severe chronic obstructive pulmonary disease with hypoxemia
13. Active bacterial, viral of fungal infection requiring systemic therapy
14. Concurrent thrombohemolytic disease
15. HIV positivity
16. HBV positivity
17. Positive serology for HBV (occult carriers: AntiHBc+, HbsAg-, AntiHbs+/-) with positive HBV-DNA test
18. HCV positivity in presence of replication marks (HCV+, CRP+, AST 1,5-2 times normal ranges)
19. CNS localization of disease
20. Prior (during last 3 years) or concurrent malignancy except adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix or early stage prostate cancer not requiring systemic therapy, or early breast cancer treated with surgery alone. Any other co.existing medical condition that would preclude study therapy administration
21. Pregnancy or breast-feeding women
22. Inability of the patient to give her/his informed consent
23. Known hypersensitivity or anaphylactic reaction to murine antibodies or proteins

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 399 (Estimated)
Dates: Start 2006-01; Primary Completion 2011-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the activity of arms "R-MegaCHOP14/R-CHOP14 + R-MAD+BEAM and ASCT" and "R-MegaCHOP14/R-CHOP14" in terms of 2-years Failure Free Survival (FFS). | 2 years

SECONDARY OUTCOMES:
To evaluate the activity of arms "R-MegaCHOP14/R-CHOP14 + R-MAD+BEAM and ASCT" and "R-MegaCHOP14/R-CHOP14" in terms of 3-years Overall Survival (OS). | 3 years
To evaluate the efficacy of two different dose-dense + Rituximab chemotherapy regimens in term of 2-years Failure Free Survival (FFS). | 2 years
To evaluate the activity of the first four courses of two different dose dense + Rituximab chemotherapy regimens (standard dose R-CHOP14 or intensified dose R-MegaCHOP14) in terms of Overall Response Rate (ORR) and Complete Remission (RC). | 2 years
To evaluate the efficacy of the four different induction arms in terms of 2-years FFS (exploratory analysis). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Principal Investigator — S.C. Ematologia II - OSP.S. GIOV.BATTISTA MOLINETTE - TORINO (TO) -
Locations (75):
- Italy (75):
  - Ospedale Umberto I - DH Oncoematologico, Nocera Inferiore, Salerno
  - Ospedale Civile Umberto I, Mestre, Venezia
  - Osp. Calvi, Noale, Mirano, Venezia
  - Az. Osp. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Cardinal Massaia, Asti
  - Centro di Riferimento Oncologico, Aviano - PN
  - Azienda Ospedale Policlinico Consorziale, Bari
  - IRCC Istituto tumori Ematologia, Bari
  - Osp. Degli Infermi, Biella
  - Ospedale Policlinico S. Orsola Malpighi, Bologna
  - Spedali Civili, Brescia
  - UTMO Ematologia Università Spedali Civili, Brescia
  - Stabilimento "Perrino", Brindisi
  - Ospedale di Circolo, Busto Arsizio - VA
  - Ospedale Armando Businco, Cagliari
  - Università Cattolica del Sacro Cuore, Campobasso
  - IRCC, Candiolo (TO)
  - Ospedale Pugliese, Catanzaro
  - Ospedale Bufalini, Cesena - FC
  - Stabilimento Ospedaliero, Ciriè - to
  - Ospedale Generale di Zona, Civitanova Marche (MC)
  - Presidio Ospedaliero Annunziata, Cosenza
  - Istituti Ospitalieri, Cremona
  - Az. Ospedaliero Universitaria Careggi, Florence
  - Stabilimento Forlì, Forlì
  - Azienda Universitaria San Martino, Genova
  - A.S.L. 9, Ivrea
  - Ospedale Felettino, La Spezia
  - Istituto Vito Fazzi, Lecce
  - Azienda Ospedaliera Papardo, Messina
  - Azienda Ospedaliero Universitaria Policlinico Gaetano Martino, Messina
  - Istituto Europeo di Oncologia, Milan
  - Osp. San Carlo Borromeo, Milan
  - Ospedale Cà Grande - Niguarda, Milan
  - Ospedale Fatebenefratelli, Milan
  - Presidio Osp. Maggiore Policlinico, Milan
  - Azienda Ospedaliera Policlinico, Modena
  - Ospedale S. Gerardo, Monza
  - Università degli Studi Federico II, Napoli
  - Osp. Maggiore Della Carità, Novara
  - Ospedale S. Francesco, Nuoro
  - Ospedale San Luigi, Orbassano (TO)
  - Azienda Ospedaliera, Padua
  - Università degli Studi, Parma
  - Fond. Maugeri - Centro medico, Pavia
  - Ospedale Policlinico San Matteo, Pavia
  - Ospedale di Piacenza, Piacenza
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Ospedale San Carlo, Potenza
  - Ospedale Santa Maria delle Croci, Ravenna
  - Ospedale Bianchi Melacrino Morelli, Reggio Calabria
  - Ospedale Santa Maria Nuova, Reggio Emilia
  - Ospedale Oncologico Regionale, Rionero in Vulture (PZ)
  - Istituto Regina Elena, Roma
  - Ospedale S. Eugenio, Roma
  - Policlinico Universitario A. Gemelli, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - Università degli Studi di Roma "La Sapienza", Roma
  - Università degli Studi di Roma 'Tor Vergata', Roma
  - Ospedale di Ronciglione, Ronciglione (VT)
  - Istituto Clinico Humanitas, Rozzano - MI
  - Casa Sollievo della Sofferenza, San Giovanni Rotondo (FG)
  - Ospedale SS.Annunziata, Sassari
  - Spedali Riuniti, Siena
  - Ospedale Morelli, Sondalo
  - Stabilimento SS. Annunziata, Taranto
  - Azienda Ospedaliera di Perugia, Terni
  - Osp. S. Giovanni Battista "Molinette", Torino
  - Ospedale Ca Focello, Treviso
  - Presidio Ospedaliero di Vittorio Veneto, Treviso
  - Ospedale Generale Prov. Cardinale G. Panico, Tricase (LE)
  - Policlinico Universitario, Udine
  - Osp. di Circolo e Fondazione Macchi, Varese
  - Stabilimento Ospedaliero, Verbania
  - Osp. Sant'Andrea Divisioen di Onco-Ematologia, Vercelli

REFERENCES:
- [Derived] Derenzini E, Mazzara S, Melle F, Motta G, Fabbri M, Bruna R, Agostinelli C, Cesano A, Corsini CA, Chen N, Righi S, Sabattini E, Chiappella A, Calleri A, Fiori S, Tabanelli V, Cabras A, Pruneri G, Vitolo U, Gianni AM, Rambaldi A, Corradini P, Zinzani PL, Tarella C, Pileri S. A three-gene signature based on MYC, BCL-2 and NFKBIA improves risk stratification in diffuse large B-cell lymphoma. Haematologica. 2021 Sep 1;106(9):2405-2416. doi: 10.3324/haematol.2019.236455. PMID 32817282
- [Derived] Chiappella A, Martelli M, Angelucci E, Brusamolino E, Evangelista A, Carella AM, Stelitano C, Rossi G, Balzarotti M, Merli F, Gaidano G, Pavone V, Rigacci L, Zaja F, D'Arco A, Cascavilla N, Russo E, Castellino A, Gotti M, Congiu AG, Cabras MG, Tucci A, Agostinelli C, Ciccone G, Pileri SA, Vitolo U. Rituximab-dose-dense chemotherapy with or without high-dose chemotherapy plus autologous stem-cell transplantation in high-risk diffuse large B-cell lymphoma (DLCL04): final results of a multicentre, open-label, randomised, controlled, phase 3 study. Lancet Oncol. 2017 Aug;18(8):1076-1088. doi: 10.1016/S1470-2045(17)30444-8. Epub 2017 Jun 28. PMID 28668386